CLINICAL TRIAL: NCT00084292
Title: International Pediatric Stroke Study
Brief Title: Database for Stroke in Infants and Children: the International Pediatric Stroke Study
Acronym: IPSS
Status: Recruiting | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Nomazulu Dlamini, Staff Physician, Neurology, The Hospital for Sick Children
Other Study IDs: 1000070460; 04-N-0210 (Registry Identifier: IPSS); 1000070460 (Registry Identifier: The International Pediatric Stroke Study)
Record Dates: First submitted 2004-06-09; First posted 2004-06-10 (Estimated); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Cerebrovascular Accident; Focal Infarct
Keywords: Ischemia; Pediatric; Etiology; Treatment; Outcome; Childhood Stroke; Pediatric Stroke; Ischemic Stroke; Spastic Hemiplegia; Hemiplegic cerebral palsy; Neonatal Stroke; Neuroimaging; Arteriopathy; Hemorrhagic
MeSH Terms: conditions — Stroke; Ischemia; Ischemic Stroke; Hemiplegia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | US Export: No

SUMMARY:
The International Pediatric Stroke Study (IPSS) was established in 2003 as a multi-center, multi-national clinical research registry. Over the years, it has grown to become a highly successful study vehicle for pediatric stroke research across over 100 institutions worldwide. Today, The IPSS continues to serve as the global clinical data and imaging core for multi-disciplinary pediatric experts who perform international collaborative research to better understand, prevent, and improve outcomes in pediatric stroke. The robust dataset and cohesive network enable high caliber and ground-breaking research in the field.

Participating sites enroll neonates or children who have had an ischemic or hemorrhagic stroke, or may be at high risk of having a stroke. Participants have their medical and research records reviewed for information about their stroke and abstracted into a secure electronic database called REDCap, which is hosted at SickKids in Toronto Canada. The IPSS also provides an attractive imaging platform (through the Stroke Imaging Lab for Children, SILC, housed at SickKids) for sites to share clinically acquired brain images that will complement the clinical dataset. The clinical and imaging datasets will improve our understanding of the processes underlying plasticity and recovery in childhood stroke.

DETAILED DESCRIPTION:
OBJECTIVES: This is the first multi-center, multi-national study of children with stroke. It seeks to build a network of investigators and high-quality disease dataset to enable population-based studies, natural history studies, and clinical trials to improve the care of children with stroke.

STUDY POPULATION: Infants and children with ischemic stroke (arterial ischemic stroke and cerebral sinovenous thrombosis), hemorrhagic stroke or those at high risk (e.g. arteriopathies like moyamoya).

DESIGN: This study includes a data collection component and collaborative process. Our network of over 150 investigators prospectively collect data on neonates or children with a diagnosis of stroke made after January 2003. Data on stroke diagnosis, etiology, treatment and outcomes are collected and entered into a secure web system, REDCap. Neuro-imaging data from the index event and a series of follow-up time points are captured and stored in the SILC-IPSS data repository.

OUTCOME MEASURES: This study will quantify outcome event rates (initial stroke characteristics, recurrent stroke, mortality, neurologic deficits), which can be used in designing future intervention studies and determining sample sizes. Analysis will be primarily descriptive. Participating investigators submit investigator-initiated research proposals or grants with a specific focus, leveraging the clinical and imaging dataset.

ELIGIBILITY:
Inclusion Criteria:

This registry will include all children from birth to 18 years of age who are diagnosed with stroke or a condition/disease (as defined below) that put them at high risk of stroke after Jan 1,2003 at one of the IPSS participating sites.

This registry will include children diagnosed with below stroke types:

* Arterial Ischemic Stroke (AIS),
* Cerebral Sinovenous Thrombosis (CSVT),
* AIS and CSVT
* Presume Preinatal Ischemic Stroke (PPIS)
* Children diagnosed with hemorrhagic stroke

Children at high risk of stroke include:

* Those diagnosed with arteriopathy, arteritis/vasculitis, moyamoya, dissection, sickle cell related infarcts).
* Brain arteriovenous malformations

Exclusion Criteria:

* Premature children diagnosed with AIS.
* Premature children diagnosed with PPIS
* Children diagnosed with TIA (Transient Ischemic Attack)
* Brain hemorrhage secondary to trauma
* Refusal to provide consent for participation

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Neonates (<28 days) and children (>29 days) to 18 years old with arterial ischemic stroke, cerebral sinovenous thrombosis, hemorrhagic stroke or at high risk of stroke
Sampling Method: Probability Sample
Enrollment: 12000 (Estimated)
Dates: Start 2003-01 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Change from Pediatric Stroke Outcome Measure at 3 months. | 3-12 months post-stroke
  The Pediatric Stroke Outcome Measure (PSOM) was developed out of a need for an objective, standardized outcome measures for children with acute, unilateral focal CNS such as cerebral infarction. The goal was to develop an assessment measure that defines clinically and functionally relevant outcome in pediatric stroke. This measure was designed for and tested in children with arterial ischemic stroke or cerebral sinovenous thrombosis.
Recovery and Recurrence Questionnaire | 3-12 months post-stroke
  The Recurrence and Recovery Questionnaire (RRQ) was developed by converting the Pediatric Stroke Outcome Measure (PSOM) into a questionnaire for patient/parent telephone interview. The agreement and consistency of the PSOM and RRQ was then assessed, and validated. The RRQ captures the same 5 sub-domains as the PSOM in the event a patient cannot return to clinic for a follow-up visit and can be used as a measure of recovery post-stroke.
King's Outcome Scale for Childhood Head Injury (KOSCHI) | 3-12 months post-stroke
  The KOSCHI is a standardized outcome measure and was developed as a pediatric adaptation of the original adult Glasgow Outcome Scale. It is a widely used outcome measure post neurological injury in children and have been used in previous pediatric stroke research. The KOSCHI can be completed through chart review of clinical or progress notes.
modified Rankin Scale (mRS) | 3-12 months post-stroke
  The modified Rankin Scale is a standardized outcome measure that captures the degree of disability in patients who have had a stroke. It is widely used in previous pediatric stroke research to assess global neurological impairment following stroke in children. It is a single-item scale and can be completed through chart review of clinical or progress notes.

SECONDARY OUTCOMES:
Investigator-Initiated Research Studies | As proposed
  Participating in the IPSS gives investigators permission to conduct multi-site research studies, in accordance with the Publications Committee policy. Manuscripts published to date can be accessed through IPSS Central (ipss.research@sickkids.ca).

CONTACTS AND LOCATIONS:
Overall Officials: Nomazulu Dlamini, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- Hospital For Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lynch JK, Hirtz DG, DeVeber G, Nelson KB. Report of the National Institute of Neurological Disorders and Stroke workshop on perinatal and childhood stroke. Pediatrics. 2002 Jan;109(1):116-23. doi: 10.1542/peds.109.1.116. PMID 11773550
- [Background] deVeber GA, MacGregor D, Curtis R, Mayank S. Neurologic outcome in survivors of childhood arterial ischemic stroke and sinovenous thrombosis. J Child Neurol. 2000 May;15(5):316-24. doi: 10.1177/088307380001500508. PMID 10830198
- [Background] deVeber G, Andrew M, Adams C, Bjornson B, Booth F, Buckley DJ, Camfield CS, David M, Humphreys P, Langevin P, MacDonald EA, Gillett J, Meaney B, Shevell M, Sinclair DB, Yager J; Canadian Pediatric Ischemic Stroke Study Group. Cerebral sinovenous thrombosis in children. N Engl J Med. 2001 Aug 9;345(6):417-23. doi: 10.1056/NEJM200108093450604. PMID 11496852
- [Background] Golomb MR, Fullerton HJ, Nowak-Gottl U, Deveber G; International Pediatric Stroke Study Group. Male predominance in childhood ischemic stroke: findings from the international pediatric stroke study. Stroke. 2009 Jan;40(1):52-7. doi: 10.1161/STROKEAHA.108.521203. Epub 2008 Sep 11. PMID 18787197